CLINICAL TRIAL: NCT02673008
Title: Minimal Residual Disease-directed Donor Lymphocyte Infusion for Reduce of Relapse After Allogenetic Hematopoietic Stem Cell Transplantation
Brief Title: MRD-directed Donor Lymphocyte Infusion for Reduce of Relapse After Allo-HSCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MRD-directed DLI-2016
Record Dates: First submitted 2016-01-23; First posted 2016-02-03 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2016-01

CONDITIONS: Minimal Residual Disease; Donor Lymphocyte Infusion; Hematopoietic Stem Cell Transplantation; Relapse
MeSH Terms: conditions — Neoplasm, Residual; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD-directed DLI (Experimental): For patients with MRD+ and without grade II/>II aGVHD by day +60 post-transplantation, DLI was given once by day +60 and was then administered based on MRD and GVHD status. If patients were MRD negative, DLI was not given again; if patients were MRD positive and without GVHD, DLI was given monthly until GVHD occurred or MRD became negative or for a total of four times. For patients with NR or PR pre-transplantation and with MRD negative by day +60 post-transplantation, DLI was given once by day +90 regardless of MRD, and was then administered when MRD became positive. For patients with CR pre-transplantation and with MRD negative post-transplantation, DLI was not given unless MRD became positive.
  Interventions: Biological: donor lymphocyte infusion

INTERVENTIONS:
Biological: donor lymphocyte infusion — DLI was administered at a median dose of 1.0 (range 0.7-1.4) ×10*8 mononuclear cells/kg.

SUMMARY:
Allogeneic hematopoietic cell transplantation (Allo-HSCT) is an effective therapy for acute leukemia, but relapse remains an important problem. Therapy options for relapse include stopping immune suppression, re-induction of chemotherapy, donor lymphocyte infusion (DLI), and another transplantation used alone or in combination. However, the efficacy of these interventions is limited. One approach to the relapse problem is to intervene before hematologic or pathologic relapse occurs based on minimal residual disease (MRD). In this study, the efficacy of MRD-directed DLI on transplantation outcomes will be evaluated in patients with acute leukemia receiving allo-HSCT.

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (Allo-HSCT) is an effective therapy for acute leukemia, but relapse remains an important problem. Therapy options for relapse include stopping immune suppression, re-induction of chemotherapy, donor lymphocyte infusion (DLI), and another transplantation used alone or in combination. However, the efficacy of these interventions is limited. One approach to the relapse problem is to intervene before hematologic or pathologic relapse occurs based on minimal residual disease (MRD) using immune or molecular techniques.DLI is an effective post-transplantation therapy for prophylaxis of leukemia relapse, but is associated with a substantial risk of GVHD. Whether MRD-directed DLI could improve outcomes remains unclear. In this study, the efficacy of MRD-directed DLI on transplantation outcomes will be evaluated in patients with acute leukemia receiving allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute leukemia
* receiving allo-HSCT

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10-25 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
relapse rate | 1 year

SECONDARY OUTCOMES:
overall survival | 1 year
disease-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan CH, Liu DH, Liu KY, Xu LP, Liu YR, Chen H, Han W, Wang Y, Qin YZ, Huang XJ. Risk stratification-directed donor lymphocyte infusion could reduce relapse of standard-risk acute leukemia patients after allogeneic hematopoietic stem cell transplantation. Blood. 2012 Apr 5;119(14):3256-62. doi: 10.1182/blood-2011-09-380386. Epub 2012 Feb 14. PMID 22337715
- [Derived] Fan M, Wang Y, Lin R, Lin T, Huang F, Fan Z, Xu Y, Yang T, Xu N, Shi P, Nie D, Lin D, Jiang Z, Wang S, Sun J, Huang X, Liu Q, Xuan L. Haploidentical transplantation has a superior graft-versus-leukemia effect than HLA-matched sibling transplantation for Ph- high-risk B-cell acute lymphoblastic leukemia. Chin Med J (Engl). 2022 Apr 20;135(8):930-939. doi: 10.1097/CM9.0000000000001852. PMID 35467818
- [Derived] Yu S, Huang F, Fan Z, Xuan L, Nie D, Xu Y, Yang T, Wang S, Jiang Z, Xu N, Lin R, Ye J, Lin D, Sun J, Huang X, Wang Y, Liu Q. Haploidentical versus HLA-matched sibling transplantation for refractory acute leukemia undergoing sequential intensified conditioning followed by DLI: an analysis from two prospective data. J Hematol Oncol. 2020 Mar 12;13(1):18. doi: 10.1186/s13045-020-00859-5. PMID 32164760